CLINICAL TRIAL: NCT03189862
Title: A PATH (Promoting Activity and Trajectories of Health) for Children
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Leah Robinson, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00133319; 1R01HL132979-01 (NIH)
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Motor Performance; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHAMP (Experimental): CHAMP, is a mastery climate motor skills interventions, that provides children the opportunity to establish behaviors that reinforces decision-making while participating in a variety of challenging movement & physical activity tasks. Duration of CHAMP is 30 min/day 4 days/week for 30 weeks. CHAMP consist of a) a 2-3 min of motor skill introductory activity that includes a group motor activity, the teaches the lesson, includes a demonstration, and understanding of developmentally appropriate learning clues b) 25 min of motor skill instruction & practice where preschoolers engage in 3-4 motor activity stations that align with the TARGET structures c) & 2-3 min motor skill closure activity that involves a review of the lesson & critical elements.
  Interventions: Behavioral: Motor Skills Intervention
- Control - Free Play (No Intervention): The control/free play condition will be the preschools typical activity programs (i.e., outdoor/indoor recess) and will be implemented according to the existing procedures within the preschool centers. The centers outdoor program consist of outdoor free-play activity on a large playground area with a variety of play structures (swings, slides, ladders) that promote gross movement and activity in preschoolers. For the control condition, there will be no planned instruction nor activities provided by the classroom teachers.

INTERVENTIONS:
Behavioral: Motor Skills Intervention — The behavioral motor skills intervention (CHAMP) is an intervention strategy that uniquely addresses differences in children's developmental levels on an individualized basis. CHAMP does not equate to a "one size fits all" approach. Children will be in an environment that promotes opportunities for them to develop improvements in motor skills based on their specific individual needs and choices. The CHAMP intervention promotes a mastery climate that allows each individual child to be successful and learn while promoting intrinsic motivation and autonomy. CHAMP will be implemented 4x/week for 30 minutes across ≈30 weeks for ≈3000 minutes of intervention time.
  Arms: CHAMP

SUMMARY:
Physical inactivity in children is a major public health risk factor and a health objective for the nation. This study aims to investigate the short- and long-term effects of a movement and physical activity program - the Children Health and Motor Programs (CHAMP) on motor competence, perceived motor competence, and physical activity. A secondary aim of this project (i.e., Science of Behavior Change Administrative Supplement) is to examine the immediate (pre- to post-test) effects of the CHAMP intervention on self-regulation and associations between self-regulation and changes in motor competence, perceived motor competence, and physical activity. The long term goal is to provide evidence-based movement experiences during the early childhood years that promote and contribute to overall healthy growth and development.

DETAILED DESCRIPTION:
Ethnic-minorities and low income children engage in less physical activity (PA)1 and, as a result, have an increased risk of cardiovascular disease. Promoting health-enhancing and sustainable PA levels across childhood and adolescence in low income and minority populations provides important health benefits. However, most PA interventions in children have not led to long-term, sustainable PA behavior. We propose a potential limitation in PA interventions has been the lack of focus on critical developmental processes (i.e., motor development and psychological constructs including perceived competence) that are established correlates of PA and may strongly impact the long-term sustainability of children's PA behaviors.

Co-investigator, Stodden et al. proposed a developmental model hypothesizing mechanisms that promote positive longitudinal change in PA from early (≈3 yrs) to late childhood (≈12 yrs). In this model, a causal pathway that impacts PA is the development of motor competence (MC, i.e., coordination and control of human movement) and perceived motor competence (PMC; i.e., perceptions of movement capabilities). PMC is directly linked to MC and influences PA as it mediates the relationship between MC and PA across childhood. Empirical evidence supports the model's hypotheses showing that MC, PMC, and PA are positively related across childhood. Principal Investigator, Robinson found that children as early as 3 yrs old demonstrate positive associations among MC, PMC, and PA, which suggests early childhood is an optimal time to promote positive MC and PMC in order to decrease the risk of developing unhealthy PA habits.

Robinson has conceptualized and tested a theoretically grounded intervention (the Children's Health Activity Motor Program; CHAMP), which aligns with tenets of the Stodden et al. model by focusing on improving MC and PMC. Studies by the PI show highly impactful results on MC and PMC. CHAMP produced strong increases in MC (improvement to the 70th%tile, up from the 15th%tile) and PMC (30% improvement) over a 9-week intervention and results were sustained following a 12-week retention. During the 30-min intervention, CHAMP participants engaged in more PA (i.e., 50% more time) compared to children in the control.13 While these intervention results are very encouraging, there is a need to examine the long-term effects of the intervention on MC and PMC and whether improvements lead to sustained PA. To date, there have been no large-scale treatment studies that have examined the long-term effects of a MC and PA-based intervention on MC, PMC, and PA in young children.

This proposed study will address these gaps utilizing a cluster randomized control trial. The CHAMP intervention will be implemented in a high minority and low-income population, namely Head Start preschoolers (N = 300; 3.5-5 yrs old), with a 3-year follow-up to examine the immediate (pre- to post-test) and sustained (across middle childhood) impact on MC, PMC, and daily PA. 30 classes of preschool children will be randomly assigned to either the treatment (CHAMP, n = 15) or control (normal preschool free-play/recess, n = 15) conditions. The CHAMP intervention will be implemented for 30 minutes/day, 4 days/week, for 30 weeks (dose of 3000 minutes). Measurements of MC (product and process), PMC (via self-perceptions of MC), and PA (via accelerometry), will occur at baseline (month 0), post-intervention (month 9), and follow-up at May of Year 2, 3, and 4. The specific aims of this study are to:

Aim 1: Examine the immediate post-intervention effect of CHAMP (compared to control participants) on MC, PMC, and PA in preschool-age children.

Aim 2: Assess the sustainable effect of CHAMP (compared to control participants) on MC, PMC, and PA across middle childhood.

Aim 3: Examine and compare the immediate and long-term mediating effect of PMC on the relationship between MC and PA in preschool-age children in the CHAMP and control.

IMPACT: Positive findings will support the development of early childhood education MC and PA programs that promote positive and sustainable PA behaviors that contribute to healthy growth and development.

ELIGIBILITY:
Inclusion Criteria:

1. Recruitment is limited to two specific schools located in the Detroit Metro area.
2. Participants must be in the last year of preschool entering Kindergarten the next academic year is eligible to to participate in this study.

Exclusion Criteria:

1. Any preschooler with a severe developmental, cognitive, and/or physical disability as noted by school records is eligible to participate in this study but data will not be collected.

Ages: 42 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 299 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah E Robinson, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson LE. Effect of a mastery climate motor program on object control skills and perceived physical competence in preschoolers. Res Q Exerc Sport. 2011 Jun;82(2):355-9. doi: 10.1080/02701367.2011.10599764. No abstract available. PMID 21699116
- [Background] Robinson LE, Rudisill ME, Goodway JD. Instructional climates in preschool children who are at-risk. Part II: perceived physical competence. Res Q Exerc Sport. 2009 Sep;80(3):543-51. doi: 10.1080/02701367.2009.10599592. PMID 19791640
- [Background] Robinson LE. The relationship between perceived physical competence and fundamental motor skills in preschool children. Child Care Health Dev. 2011 Jul;37(4):589-96. doi: 10.1111/j.1365-2214.2010.01187.x. Epub 2010 Dec 9. PMID 21143273
- [Background] Robinson LE, Goodway JD. Instructional climates in preschool children who are at-risk. Part I: object-control skill development. Res Q Exerc Sport. 2009 Sep;80(3):533-42. doi: 10.1080/02701367.2009.10599591. PMID 19791639
- [Background] Ulrich DA. Test of gross motor development-3. Austin, TX: Prod-Ed; 2015.
- [Background] Stodden DF, Langendorfer SJ, Fleisig GS, Andrews JR. Kinematic constraints associated with the acquisition of overarm throwing part I: step and trunk actions. Res Q Exerc Sport. 2006 Dec;77(4):417-27. doi: 10.1080/02701367.2006.10599377. PMID 17243217
- [Background] Stodden DF, Langendorfer SJ, Fleisig GS, Andrews JR. Kinematic constraints associated with the acquisition of overarm throwing part II: upper extremity actions. Res Q Exerc Sport. 2006 Dec;77(4):428-36. doi: 10.1080/02701367.2006.10599378. PMID 17243218
- [Background] Harter S, Pike R. The pictorial scale of perceived competence and social acceptance for young children. Child Dev. 1984 Dec;55(6):1969-82. PMID 6525886
- [Background] Harter S. Manual for the Self-Perception Profile for Children. Denver, CO: University of Denver; 1985.
- [Background] Trost SG, McIver KL, Pate RR. Conducting accelerometer-based activity assessments in field-based research. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S531-43. doi: 10.1249/01.mss.0000185657.86065.98. PMID 16294116
- [Background] Choi L, Liu Z, Matthews CE, Buchowski MS. Validation of accelerometer wear and nonwear time classification algorithm. Med Sci Sports Exerc. 2011 Feb;43(2):357-64. doi: 10.1249/MSS.0b013e3181ed61a3. PMID 20581716
- [Background] Willoughby M, Blair C. Test-retest reliability of a new executive function battery for use in early childhood. Child Neuropsychol. 2011;17(6):564-79. doi: 10.1080/09297049.2011.554390. Epub 2011 Jun 30. PMID 21714751
- [Background] Raver CC, Jones SM, Li-Grining C, Zhai F, Bub K, Pressler E. CSRP's Impact on low-income preschoolers' preacademic skills: self-regulation as a mediating mechanism. Child Dev. 2011 Jan-Feb;82(1):362-78. doi: 10.1111/j.1467-8624.2010.01561.x. PMID 21291447
- [Derived] Wood AP, Palmer KK, Ouyang Z, Wang LU, Robinson LE. Developmental Changes in Motor Competence: The Influence of Physical Activity and BMI Percentile. Med Sci Sports Exerc. 2025 Dec 1;57(12):2690-2696. doi: 10.1249/MSS.0000000000003805. Epub 2025 Jul 3. PMID 40605193
- [Derived] Robinson LE, Palmer KK, Wang L, Scott-Andrews KQ, Chinn KM, Sur I, Wengrovius C, Meng E, Veldman SLC, Miller AL. Protocol for a cluster randomized clinical trial of a mastery-climate motor skills intervention, Children's Health Activity and Motor Program (CHAMP), on self-regulation in preschoolers. PLoS One. 2023 Mar 9;18(3):e0282199. doi: 10.1371/journal.pone.0282199. eCollection 2023. PMID 36893091
- [Derived] Robinson LE, Wang L, Colabianchi N, Stodden DF, Ulrich D. Protocol for a two-cohort randomized cluster clinical trial of a motor skills intervention: The Promoting Activity and Trajectories of Health (PATH) Study. BMJ Open. 2020 Jun 11;10(6):e037497. doi: 10.1136/bmjopen-2020-037497. PMID 32532781

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHAMP | Control - Free Play
Started | 153 | 146
Completed | 98 | 84
Not Completed | 55 | 62
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 54 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHAMP | Control - Free Play | Total
Number analyzed (Participants) | 153 | 146 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 153 | 146 | 299
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 52.5 (3.42) | 53.5 (3.99) | 53.00 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 72 | 158
  Male | 67 | 74 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 134 | 122 | 256
  Unknown or Not Reported | 15 | 16 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 96 | 90 | 186
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 33 | 32 | 65
Region of Enrollment [Number; unit: participants]
  United States | 153 | 146 | 299

OUTCOME MEASURES:

1. Primary Outcome: Motor Competence - Process Measures
Description: Motor competence process measures will be scored using the Test of Gross Motor Development-3rd Edition; scores for the two subscales - locomotor (score range: 0-46) & object-control (score range: 0-54) will be reported as raw scores for each skill & an overall score total MC score which is created by summing the subscales( score range: 0 (low motor competence) - 100 (high motor competence)). Locomotor, object control, and total raw scores will be used for data analyses when appropriate. All scores are interpreted as a higher score indicating better outcomes.
Time Frame: Baseline (Month 0), post-intervention (month 9)
Population: We had three fewer children complete locomotor skills at post-intervention due to absence on a testing day.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 144 | 132
score on a scale
  Locomotor Baseline (Month 0) | 14.24 (6.09) | 14.35 (5.98)
  Locomotor Post-Intervention (Month 9): number analyzed (Participants) | 144 | 129
  Locomotor Post-Intervention (Month 9) | 22.03 (6.98) | 17.26 (6.35)
  Ball Skills Baseline (Month 0) | 15.32 (7.15) | 15.27 (7.15)
  Ball Skills Post-Intervention (Month 9): number analyzed (Participants) | 144 | 129
  Ball Skills Post-Intervention (Month 9) | 23.97 (8.00) | 18.16 (8.10)
  Total Baseline (Month 0) | 29.57 (11.21) | 29.62 (11.37)
  Total Post-Intervention (month 9) | 45.99 (12.64) | 35.42 (12.09)

2. Primary Outcome: Physical Activity
Description: ActiGraph GTX3+ tri-axial accelerometer will be used to measure the frequency, intensity and duration of PA among children at school and in free-living settings. Participants will be asked to wear the same accelerometer for 7 full days (5 week and 2 weekend days). Data will be collected at 80 hz. Cut points from a study in preschoolers by Butte et al will be applied to activity counts. This study utilized information from all three axes (versus just the vertical axis) thus time spent in sedentary, light, moderate, and vigorous categories will be defined as vector magnitudes of up to 819 (sedentary), 3907 (light), 6111 (moderate) and above 6112 for vigorous activity. The outcome will be minutes of moderate-to-vigorous PA per day, greater than 6111 activity counts.
Time Frame: Baseline (Month 0), post-intervention (month 9)
Population: Smaller population here due to non-compliance with accelerometer wear protocols. Children had to wear the device for 7 consecutive days and have 4 valid wear days (3 weekdays and 1 weekend day) to be included in final analyses.
Measure: Mean (Standard Deviation); unit: minutes of moderate-to-vigorous PA/day
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 103 | 107
minutes of moderate-to-vigorous PA/day
  PA Baseline (month 0) | 66.97 (21.08) | 67.2 (24.75)
  PA Post-Intervention (month 9) | 74.41 (22.26) | 82.74 (29.53)

3. Primary Outcome: Motor Competence - Product Measure
Description: Motor competence product measures will consist of 1) kick & throw velocity, catching %; hop & jump distance & running speed. Product scores will vary for each participant (i.e., kick and throw velocity - faster score is an indicator of MC, number of successful catches out of 5 attempts - more catches indicator of MC, hop and jump distance and running speed; greater distance & speed is a better indicator of MC. Catching % will not be calculated into the motor competence score due to updates in the literature regarding this specific outcome. All scores are standardized (z-scores, m=0, SD=1) and summed to get a composite for ball skills (z-kick velocity + z-throw velocity), locomotor skills (z-run speed + z-hop speed, + z-jump distance), and total (all summed). A higher score reflects better competence.
Time Frame: Baseline (Month 0), post-intervention (month 9)
Measure: Mean (Standard Deviation); unit: summed z-scores
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 134 | 142
summed z-scores
  Locomotor Baseline (month 0) | -1.50 (2.13) | -1.61 (2.29)
  Locomotor Post-Intervention (month 9) | 0.25 (2.05) | -0.31 (2.26)
  Ball Skills Baseline (Month 0) | -0.90 (1.49) | -0.81 (1.57)
  Ball Skills post-intervention (month 9) | 0.25 (2.05) | -0.01 (1.69)
  Total Baseline (month 0) | -2.39 (3.18) | -2.42 (3.46)
  Total Post-Intervention (month 9) | 0.15 (3.06) | -0.31 (3.48)

4. Secondary Outcome: Duration of Changes in Motor Competence - Process Measures
Description: Motor competence process measures will be scored using the Test of Gross Motor Development-3rd Edition; scores for the two subscales - locomotor (score range: 0-46) & object-control (score range: 0-54) will be reported as raw scores for each skill & an overall score total MC score which is created by summing the subscales( score range: 0 (low motor competence) - 100 (high motor competence)). Locomotor, object control, and total raw scores will be used for data analyses when appropriate. All scores are interpreted as a higher score indicating better outcomes.
  Due to the covid-19 pandemic, data was only collected at the follow-up period in Year 2 (year 3 and 4 was not collected)
Time Frame: Follow-up measurements at year 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 98 | 82
score on a scale
  Locomotor | 21.09 (5.77) | 18.50 (5.98)
  Ball Skills | 22.67 (7.71) | 19.25 (7.27)
  Total | 43.77 (11.43) | 37.66 (11.51)

5. Secondary Outcome: Duration of Change in Physical Activity
Description: ActiGraph GTX3+ tri-axial accelerometer will be used to measure the frequency, intensity and duration of PA among children at school and in free-living settings. Participants will be asked to wear the same accelerometer for 7 full days (5 week and 2 weekend days). Data will be collected at 80 hz. Cut points from a study in preschoolers by Butte et al will be applied to activity counts. This study utilized information from all three axes (versus just the vertical axis) thus time spent in sedentary, light, moderate, and vigorous categories will be defined as vector magnitudes of up to 819 (sedentary), 3907 (light), 6111 (moderate) and above 6112 for vigorous activity. The outcome will be minutes of moderate-to-vigorous PA per day, greater than 6111 activity counts. More minutes of MVPA is better. Due to the covid-19 pandemic, data was only collected at the follow-up period in Year 2 (year 3 and 4 was not collected)
Time Frame: Follow-up measurements at year 2
Measure: Mean (Standard Deviation); unit: minutes of moderate-to-vigorous PA/day
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 78 | 62
minutes of moderate-to-vigorous PA/day | 73.26 (22.72) | 86.68 (36.56)

6. Secondary Outcome: Perceived Motor Competence (Global)
Description: Will be assessed with the Harter & Pike Pictorial Scale of PMC and Social Acceptance (PSPCSA). The PSPCSA will measure the child's global perceived physical competence. The PSPCSA physical competence subscale consists of six items that are presented in pictures and each child will select a picture that is more like them. The six items included are swinging, climbing, tying shoe laces, skipping, running, & hopping.Children will (1) select the picture that is most like them. One picture depicts a child who is skilled competent and the other shows a child who is not skilled; (2) focus on the designated picture and indicate whether they are just a "little bit" or "a lot" like that picture. Separate pictures for girls and boys will be used in accordance with the manual procedures. The range of scores for each item on the test is 1 (low competence) to 4 (high competence), and children's final score is an average scaled score across all 6 items (1= low- 4=high).
Time Frame: Baseline (Month 0), post-intervention (month 9)
Measure: Mean (Standard Deviation); unit: average scale score
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 148 | 141
average scale score
  Baseline (month 0) | 3.25 (0.61) | 3.18 (0.59)
  Post-Intervention (month 9) | 3.22 (0.63) | 3.23 (0.64)

7. Secondary Outcome: Perceived Motor Competence (Fundamental)
Description: Global perceived motor competence will be assessed with the Digital Scale of Perceived Motor Competence (DSPMC). THis video-based assessment allows children to see motor skills in action rather than a static picture. The scale is the identical layout and item structure to the PSPCSA but aligns with the 12 fundamental motor skills of the TGMD. For the assessment, the child will watch 12 sets of video pairs and select the video from each pair where the person moves most like them. One video depicts a child who is skilled and the other shows a child who is not skilled. Once children select the video where the person moved like them, they indicate whether the person in the video moved a "little bit" or "a lot" like themselves. The DSPMC yields three scores- locomotor (6 video pairs), ball skills (6 video pairs), and total (all 12 video pairs). The final score from each is an average scale score that ranges in value from 1 (low perceived competence) to 4 (high perceived competence).
Time Frame: Baseline (Month 0), post-intervention (month 9)
Measure: Mean (Standard Deviation); unit: average scale score
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 148 | 141
average scale score
  Locomotor Baseline (month 0) | 2.90 (0.45) | 2.82 (0.46)
  Locomotor Post-Intervention (month 9) | 3.13 (0.55) | 2.94 (0.46)
  Ball Skills Baseline (month 0) | 2.81 (0.48) | 2.83 (0.49)
  Ball Skills Post-Intervention (month 9) | 3.08 (0.52) | 2.92 (0.48)
  Total Baseline (month 0) | 2.86 (0.39) | 2.82 (0.40)
  Total Post-Intervention (month 9) | 3.11 (0.48) | 2.93 (0.38)

8. Secondary Outcome: Duration of Change in Perceived Motor Competence (Global)
Description: as for outcome 6
Time Frame: Follow-up measurements at year 2
Measure: Mean (Standard Deviation); unit: average scale score
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 98 | 84
average scale score | 3.38 (0.63) | 3.44 (0.51)

9. Secondary Outcome: Duration of Change in Perceived Motor Competence (Fundamental)
Description: as for outcome 7
Time Frame: Follow-up measurements at year 2
Measure: Mean (Standard Deviation); unit: average scale score
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 98 | 84
average scale score
  Locomotor (Follow Up) | 3.29 (0.53) | 3.19 (0.48)
  Ball Skill (Follow Up) | 3.19 (0.49) | 3.15 (0.44)
  Total (Follow Up) | 3.24 (0.44) | 3.17 (0.39)

10. Secondary Outcome: Cognitive Flexibility
Description: The Dimensional Change Cart Sort (DCCS) Task is a measure of cognitive flexibility. The task requires children to learn and remember a rule and apply it one way, and then apply a new rule as instructions change. Children match pictures that vary by two dimensions, shape (rabbit vs. boat) and color (brown vs. white). Children complete trials with one set of instructions, then another, and are encouraged to go as fast as they can without making mistakes. The final score was between 0-12, one point for each stimulus sorted correctly after the sort.
Time Frame: Baseline (Month 0), post-intervention (month 9)
Population: NOTE: These data were a part of a supplement and were only collected on one cohort, resulting in lower sample sizes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 68 | 46
score on a scale
  Baseline (month 0) | 2.25 (3.32) | 1.83 (3.01)
  Post-Intervention (month 9) | 4.62 (4.07) | 4.86 (3.86)

11. Secondary Outcome: Working Memory
Description: Working Memory will be assessed using a visual-spatial working memory task which requires children to accurately recall information they have seen before. Children are shown visual information (stickers on the body of a cartoon character) and next shown the character without the stickers, and asked to identify these locations after a brief retention interval. Test trials increase in difficulty (i.e., WM demand) as the task progresses. Test continues until a max. of 8 levels or failure on all 3 trials at the same level of difficulty. For working memory, more accurate responses reflect better self-regulation.WM capacity was indexed by a point score calculated as follows: beginning from Level 1, one point for each consecutive level in which at least two of the three trials were performed accurately, plus 1/3 of a point for all correct trials thereafter. Therefore, final scores are between 0-8 with higher scores reflecting better working memory.
Time Frame: Baseline (Month 0), post-intervention (month 9)
Population: NOTE: These data were a part of a supplement and were only collected on one cohort, resulting in lower sample sizes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 70 | 46
score on a scale
  Baseline (month 0) | 0.64 (0.86) | 0.63 (0.87)
  Post-Intervention (month 9) | 1.03 (1.09) | 1.02 (0.96)

12. Secondary Outcome: Behavioral Inhibition
Description: The Head-Toes-Knees-Shoulders Task (HTKS; 10 min.) will be used to measure behavioral inhibition. It reflects a child's ability to remember commands and to behaviorally inhibit a pre-potent response in favor of a less-dominant response. A child is trained to perform actions in response to an examiner's commands (e.g., "touch your toes") then asked to do the opposite (e.g., touch toes when instruction is "touch your head"). Scores across trials are summed to reflect self-regulation. The task has begins with 6 practice items and between the first and second set of items there are 5 more practice trials. The score range is 0-60; higher score equal better behavioral inhibition.
Time Frame: Baseline (Month 0), post-intervention (month 9)
Population: NOTE: These data were a part of a supplement and were only collected on one cohort, resulting in lower sample sizes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 69 | 46
score on a scale
  Baseline (month 0) | 12.13 (17.25) | 7.24 (12.18)
  Post-Intervention (month 9) | 25.31 (24.88) | 16.48 (21.39)

13. Secondary Outcome: Observed Self-Regulation
Description: Observed self-regulation will also evaluate the child ability to stay on-task during Head-Toes-Knees-Shoulders (HTKS) as an aspect of self-regulation. Child compliance and engagement will also be rated using the Child Assessor Report which has been used in prior SR trials. This 10-item questionnaire is scored on a 0-3 scale. The average scale score is taken across the 10-items, and higher score indicates better observed self-regulation behaviors.
Time Frame: Baseline (Month 0), post-intervention (month 9)
Population: NOTE: These data were a part of a supplement and were only collected on one cohort, resulting in lower sample sizes.
Measure: Mean (Standard Deviation); unit: avg scale score
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 70 | 47
avg scale score
  Baseline (month 0) | 2.48 (0.55) | 2.39 (0.47)
  Post-Intervention (month 9) | 2.48 (0.43) | 2.33 (0.62)

14. Secondary Outcome: Teacher Reported Self-Regulation
Description: Teacher-Reported. Teachers will report on child emotion regulation, another key aspect of SR at this age, using the 24-item Emotion Regulation Checklist (ERC), which generates Emotion Regulation and Negative Lability subscales. It is a 24 item, four-point Likert scale 1 = Never to 4 = Almost Always). The avg scale score is taken for both Emotional Regulation and Negative Labiltiy and a higher score indicates better emotional regulation (i.e., self-regulation behaviors).
Time Frame: Baseline (Month 0), post-intervention (month 9)
Population: NOTE: These data were a part of a supplement and were only collected on one cohort, resulting in lower sample sizes.
Measure: Mean (Standard Deviation); unit: avg scale score
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 69 | 45
avg scale score
  Emotional Reg Baseline (month 0) | 3.47 (0.46) | 3.42 (0.56)
  Emotional Regulation Post-Intervention (month 9) | 3.55 (0.44) | 3.38 (0.58)
  Neg Lability Baseline (month 0) | 1.60 (0.70) | 1.61 (0.68)
  Neg Lability Post-Intervention (month 9) | 1.52 (0.55) | 1.49 (0.51)

15. Secondary Outcome: Duration of Change Motor Competence - Product Measure
Description: as for outcome 3
Time Frame: Follow-up measurements at year 2
Measure: Mean (Standard Deviation); unit: summed z-scores
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 87 | 80
summed z-scores
  Locomotor (Follow Up) | 1.23 (2.21) | 1.15 (2.47)
  Ball Skills (Follow Up) | 0.32 (1.36) | 0.55 (1.88)
  Total (Follow Up) | 1.60 (3.11) | 1.69 (3.88)

16. Other Pre Specified Outcome: Body Mass Index
Description: Body mass index (BMI) is a weight outcome that will be collected to calibrate actigraphs and as a confounding variable. Height and weight will be used to calculate BMI. Height will be measured to the nearest unit (in centimeters) in bare feet with the child standing upright against a portable stadiometer (Charder HM200P PortStad, Taiwan ROC). Weight will be measured to the nearest unit (in kilograms) with heavy clothes removed (ie, wearing pants and shirt) using a portable electric weight scale (Seca 813; Seca North America). Body mass index (BMI) will be calculated based on age-specific and sex-specific CDC (Centers for Disease Control and Prevention) growth charts using the following formula ~ weight (kg) / [height (m)]2. BMI scores are not linear and both very high and very low BMI scores are indicative of poor health.
  Due to the covid-19 pandemic, data was only collected at the follow-up period in Year 2 (year 3 and 4 was not collected)
Time Frame: Baseline (Month 0), post-intervention (month 9), follow-up measurement at year 2
Population: Loss of sample size at follow up
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 151 | 144
kg/m^2
  Baseline | 16.44 (2.05) | 16.58 (2.04)
  Post-Intervention | 16.43 (2.06) | 16.73 (2.37)
  Follow Up: number analyzed (Participants) | 98 | 84
  Follow Up | 16.53 (1.91) | 16.70 (2.80)

17. Other Pre Specified Outcome: Waist Circumference
Description: Waist circumference is a weight outcome that will be collected as a confounding variable. The measure will be collected with the standard procedures - a non-elastic tape measure (Seca 201; Seca North America, Chino, California, USA) at the umbilicus. The measurement will be taken as the children complete a breath (ie, exhaled) to the nearest unit (in centimeters).
  Due to the covid-19 pandemic, data was only collected at the follow-up period in Year 2 (year 3 and 4 was not collected)
Time Frame: Baseline (Month 0), post-intervention (month 9), Follow-up measurement at year 2
Population: Note- change in sample size at timepoint 3 due to loss to follow up
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 152 | 143
cm
  Baseline (month 0) | 53.94 (5.55) | 54.14 (5.84)
  Post-Intervention (month 9) | 54.73 (5.02) | 55.82 (6.69)
  Follow up: number analyzed (Participants) | 98 | 83
  Follow up | 55.87 (4.88) | 56.47 (6.80)

18. Other Pre Specified Outcome: Body Fat Percentage
Description: Body fat percentage is a weight outcome that will be collected as a confounding variable. A Tanita SC-331S foot-to-foot body composition analyzer (Tanita Cooperation, Tokyo, Japan) will be used to assess bioelectrical impedance. Measurements were collected using the standard setting after manually imputing the measured height, gender, and age of the subject. The children were bare foot and wore minimal clothing and were instructed to standstill with their feet touching all four metal plates. BF% was then estimated using the in-built Tanita equations. FM (kg) was calculated as: BF% divided by 100 and then multiplied by body weight and FFM (kg) was subsequently calculated as the difference of body weight and FM. Due to the covid-19 pandemic, data was only collected at the follow-up period in Year 2 (year 3 and 4 was not collected)
Time Frame: Baseline (Month 0), post-intervention (month 9), Follow-up measurement at Year 2
Population: Due to equipment not arriving on time, we did not collect body fat on cohort one at baseline. The other change in sample size at follow-up was due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | CHAMP | Control - Free Play
Number analyzed (Participants) | 123 | 132
percentage of body fat
  Baseline (month 0): number analyzed (Participants) | 81 | 94
  Baseline (month 0) | 22.86 (5.19) | 22.08 (5.18)
  Post Intervention (month 9) | 22.13 (4.90) | 22.81 (5.09)
  Follow Up: number analyzed (Participants) | 97 | 84
  Follow Up | 21.86 (4.59) | 21.75 (5.64)

ADVERSE EVENTS:
Time Frame: Adverse events were collected across the duration of the study: baseline testing (month 0), intervention (month 1-8), post-intervention testing (month 9), and follow-up (1-year post post-intervention).
Description: Adverse events were collected through reports from research staff and included any event that had to be logged with the school front office or the IRB.
Arm/Group | CHAMP | Control - Free Play
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/146
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/146
Other Adverse Events (participants affected / at risk) | 0/153 | 0/146

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT03189862/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03189862/SAP_001.pdf
  • Informed Consent Form (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03189862/ICF_002.pdf